CLINICAL TRIAL: NCT01839708
Title: Mothers in Motion Program to Prevent Weight Gain in Overweight/Obese WIC Mothers (MIM)
Brief Title: Mothers in Motion Program to Prevent Weight Gain in WIC Mothers (MIM)
Acronym: MIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Mei-Wei Chang, Associate Professor, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1R18DK083934-01A2 (NIH)
Record Dates: First submitted 2013-02-28; First posted 2013-04-25 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-04

CONDITIONS: Overweight; Obesity
Keywords: Intervention
MeSH Terms: conditions — Overweight; Obesity | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Counseling (Experimental): Intervention group: in addition to usual WIC care, watch the DVDs at home, complete action plan worksheets, call in to moderated (MI) group discussions.
  Interventions: Behavioral: Lifestyle Counseling
- No Lifestyle Counseling (No Intervention): Comparison group: usual WIC care; read printed materials at home

INTERVENTIONS:
Behavioral: Lifestyle Counseling — The intervention will determine the differential outcomes of reading generic materials versus viewing custom DVDs containing targeted health information and discussions with MI-trained moderators on weight gain prevention.
  Other Names: Motivational Interviewing
  Arms: Lifestyle Counseling

SUMMARY:
Mothers in Motion will draw on the successes of the pilot intervention of the same name and will promote healthy lifestyle behavior changes (eating more fruits and vegetables, increasing physical activity, dealing with stress) in low-income WIC mothers of young children. The intervention group's weight change (difference between the initial enrollment and 3 months post intervention) will differ from the control group's weight change by an average of at least 2.8 pounds.

DETAILED DESCRIPTION:
Mothers in Motion will draw on the successes of the pilot intervention of the same name and will promote healthy lifestyle behavior changes (eating more fruits and vegetables, increasing physical activity, dealing with stress) in low-income WIC mothers of young children. Both treatment groups will receive usual WIC care (nutrition counseling and similar services). The control group will receive generic printed health and nutrition materials to read at their own pace if they wish. The intervention group will watch the culturally sensitive DVD chapters according to a study calendar, complete action plan worksheets, and call in to peer support group teleconferences to discuss the DVD chapter contents. The teleconferences will be led by moderators trained in motivational interviewing (MI) and group facilitation. Participants will complete phone interviews and provide body weight measurements at baseline (T1), immediately after (T2) and 3 months after (T3) the intervention time period. T3 body weight will be the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* African American or White
* Fluent in English
* 18-39 years old
* At least 6 weeks postpartum
* Body Mass Index (BMI) between 25.0 and 39.9
* Willing to provide address and up to 3 working phone numbers
* Willing to update their contact information monthly
* Willing to participate in the project for 9 months
* Willing to make 3 additional trips to WIC clinics for weight measures
* Working DVD player at home and access to a working phone.

Exclusion Criteria:

* Pregnant
* MIM Pilot study participation
* Plan to become pregnant or relocate to a location outside of study area during the trial
* Self-reported type 1 or 2 Diabetes
* Unable to walk more than 1 block without resting or shortness of breath.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 569 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Wei Chang, Ph.D, Principal Investigator — Michigan State University College of Nursing
Locations (2):
- United States (2):
  - Michigan State University, East Lansing, Michigan
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chang MW, Brown R, Nitzke S. Results and lessons learned from a prevention of weight gain program for low-income overweight and obese young mothers: Mothers In Motion. BMC Public Health. 2017 Feb 10;17(1):182. doi: 10.1186/s12889-017-4109-y. PMID 28187726
- [Derived] Chang MW, Brown R, Wegener DT. Perceived stress linking psychosocial factors and depressive symptoms in low-income mothers. BMC Public Health. 2021 Jan 6;21(1):62. doi: 10.1186/s12889-020-10118-4. PMID 33407305
- [Derived] Chang MW, Robbins LB, Ling J, Brown R, Wegener DT. Mediators affecting the association between a lifestyle behavior intervention and stress in low-income overweight or obese mothers of young children. J Health Psychol. 2021 Sep;26(10):1625-1636. doi: 10.1177/1359105319887780. Epub 2019 Nov 21. PMID 31749377
- [Derived] Chang MW, Brown R, Wegener DT, Brill S, Schaffir J, Hu J. Chaos and psychosocial health in low-income overweight or obese women. Health Psychol. 2019 Dec;38(12):1159-1167. doi: 10.1037/hea0000813. Epub 2019 Oct 3. PMID 31580130
- [Derived] Chang MW, Tan A, Schaffir J, Wegener DT. Sleep and weight loss in low-income overweight or obese postpartum women. BMC Obes. 2019 Apr 1;6:12. doi: 10.1186/s40608-019-0236-6. eCollection 2019. PMID 30984405
- [Derived] Chang MW, Nitzke S, Brown R. Mothers In Motion intervention effect on psychosocial health in young, low-income women with overweight or obesity. BMC Public Health. 2019 Jan 14;19(1):56. doi: 10.1186/s12889-019-6404-2. PMID 30642311
- [Derived] Chang MW, Brown R, Nitzke S. A Community-Based Intervention Program's Effects on Dietary Intake Behaviors. Obesity (Silver Spring). 2017 Dec;25(12):2055-2061. doi: 10.1002/oby.21862. Epub 2017 Oct 31. PMID 29086490
- [Derived] Chang MW, Hales D, Brown R, Ward D, Resnicow K, Nitzke S. Validation of PIN 3 physical activity survey in low-income overweight and obese young mothers. BMC Public Health. 2015 Feb 10;15:121. doi: 10.1186/s12889-015-1493-z. PMID 25885482
- [Derived] Chang MW, Nitzke S, Brown R, Resnicow K. A community based prevention of weight gain intervention (Mothers In Motion) among young low-income overweight and obese mothers: design and rationale. BMC Public Health. 2014 Mar 25;14:280. doi: 10.1186/1471-2458-14-280. PMID 24666633

RESULTS

PARTICIPANT FLOW:
Groups:
- No Lifestyle Counseling: Comparison group: usual WIC care; read printed materials at home
  Lifestyle Counseling: The intervention will determine the differential outcomes of reading generic materials versus viewing custom DVDs containing targeted health information and discussions with MI-trained moderators on weight gain prevention.
Period: Overall Study
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Started | 387 | 182
Completed | 311 | 115
Not Completed | 76 | 67

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling | Total
Number analyzed (Participants) | 387 | 182 | 569
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 387 | 182 | 569
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 387 | 182 | 569
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 387 | 182 | 569

OUTCOME MEASURES:

1. Primary Outcome: Measured Body Weight
Description: measured body weight in person at WIC office
Time Frame: 3 months after the 16-week intervention (T3)
Population: The inconsistent number of participants that were reported because we conducted general linear mixed model for repeated measures, which is a partial intention-to-treat analysis (ITT), adjusting baseline assessment. We chose to perform this method without any ad hoc imputation as our approach to ITT because the overall high dropout was high
Measure: Mean (Standard Error); unit: lbs
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 196 | 115
lbs | 188.3 (10.6) | 187.7 (10.6)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p > 0.05, Mixed Models Analysis

2. Secondary Outcome: T1 Fat Intake
Description: self-reported fat intake behavior using Rapid Food Screener (17 items total). Responses to each fat intake item were rated on a 5-point scale ranging from 0 (1 time or less per month) to 4 (5 or more times per week). Summed responses ranged from 0 to 68.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 387 | 182
units on a scale | 22.59 (8.81) | 21.75 (8.89)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p > 0.05, Mixed Models Analysis

3. Secondary Outcome: T1 Fruit and Vegetable Intake
Description: self-reported fruit and vegetable intake (7 items total). Responses to each fruit and vegetable intake item were rated on a 6-point scale and were rated as 0 = less than 1 time per week, 1 = once a week, 2 = 2-3 times a week, 3 = 4-6 times a week, 4 = once a day, and 5 = 2 or more times a day. Summed responses ranged from 0 to 35.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 387 | 182
units on a scale | 11.3 (4.67) | 10.89 (4.64)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p < 0.05, Mixed Models Analysis

4. Secondary Outcome: T1 Physical Activity
Description: Self-reported using the Pregnancy Infection and Nutrition 3 survey (24 items/activities). Participants reported frequency and duration (in hours) of physical activity that was done in seven categories and in the past 7 days. These categories were recreation (4 activities), indoor (5 activities) and outdoor (4 activities) household tasks, child and adult care (5 activities), transportation (2 activities) and activity at work and school (4 items). We first calculated hours spent on (frequency x duration) each activity, then sum all activities from 7 categories to create the total hours of moderate physical activity in the past 7 days (range 0 to 72 hours/past 7 days). The more hours, the more physical activity.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 387 | 182
hours | 14.720 (54.949) | 7.757 (19.723)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p > 0.05, Mixed Models Analysis

5. Secondary Outcome: T1 Stress
Description: Self-report using the Perceived Stress Scale (9 items) to measure stress perception. Participants were asked about their perception of stress in the past month. Response options were scored on a 4-point scale ranging from 1 (rarely or never) to 4 (usually or always). The overall stress score was the mean of the 9-item scores, with a higher score indicating lower stress.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 387 | 182
units on a scale | 3.28 (0.56) | 3.24 (0.51)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p < 0.05, Mixed Models Analysis

6. Secondary Outcome: T2 Fat Intake
Description: as for outcome 2
Time Frame: immediately after the 16-week intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 212 | 126
units on a scale | 17.16 (7.43) | 18.99 (10.90)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p = 0.03, Mixed Models Analysis

7. Secondary Outcome: T3 Fat Intake
Description: as for outcome 2
Time Frame: 3-month after the 16-week intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 196 | 115
units on a scale | 18.42 (8.96) | 17.22 (10.94)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p < 0.05, Mixed Models Analysis

8. Secondary Outcome: T2 Fruit and Vegetable Intake
Description: as for outcome 3
Time Frame: immediately after the 16-week intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 212 | 126
units on a scale | 11.11 (4.08) | 10.90 (4.15)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p < 0.05, Mixed Models Analysis

9. Secondary Outcome: T3 Fruit and Vegetable Intake
Description: as for outcome 3
Time Frame: 3-month after the 16-week intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 196 | 115
units on a scale | 11.77 (4.90) | 10.97 (6.01)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p < 0.05, Mixed Models Analysis

10. Secondary Outcome: T2 Physical Activity
Description: as for outcome 4
Time Frame: immediatly after the 16-week intervention
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 213 | 127
Hours | 5.389 (25.953) | 4.967 (12.290)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p < 0.05, Mixed Models Analysis

11. Secondary Outcome: T3 Physical Activity
Description: as for outcome 4
Time Frame: 3-month after the 16-week intervention
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 198 | 116
Hours | 4.417 (16.273) | 3.666 (12.000)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p < 0.05, Mixed Models Analysis

12. Secondary Outcome: T2 Stress
Description: as for outcome 5
Time Frame: immediatly after the 16-week intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 212 | 126
units on a scale | 2.56 (0.358) | 2.44 (0.356)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p < 0.05, Mixed Models Analysis

13. Secondary Outcome: T3 Stress
Description: as for outcome 5
Time Frame: 3-month after the 16-week intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 196 | 115
units on a scale | 2.55 (0.35) | 2.51 (0.356)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p < 0.05, Mixed Models Analysis

14. Secondary Outcome: Measured Body Weight
Description: measured body weight in person at WIC office
Time Frame: Immediatly after the 16-week intervention (T2)
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
Number analyzed (Participants) | 219 | 124
lbs | 188.45 (10.84) | 188.52 (10.87)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs No Lifestyle Counseling; Test type: Other; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Immediately after the 16-week intervention (T2) and 3 months after the 16-week intervention (T3)
Arm/Group | Lifestyle Counseling | No Lifestyle Counseling
All-Cause Mortality (participants affected / at risk) | 0/387 | 0/182
Serious Adverse Events (participants affected / at risk) | 0/387 | 0/182
Other Adverse Events (participants affected / at risk) | 0/387 | 0/182

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No